CLINICAL TRIAL: NCT07304869
Title: Comparison of Treatment Durations for Endodontic Procedures on Maxillary Molar Teeth Using Different Magnification Techniques
Brief Title: Treatment Durations for Endodontic Procedures
Status: Completed | Type: Observational
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Oğuz Tavşan, Assistant professor, Uşak University
Other Study IDs: 558-558-07
Record Dates: First submitted 2025-11-26; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-11

CONDITIONS: Root Canal Therapy
Keywords: root canal treatment; Dental operating microscope; dental loupes; chair time; second mesiobuccal canal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients treated under direct vision: Root canal treatment of maxillary first molar teeth performed without magnification, using direct visual inspection only.
- Patients treated using dental loupes: Root canal treatment of maxillary first molar teeth performed using 5× magnification dental loupes.
- Patients treated using a dental operating microscope: Root canal treatment of maxillary first molar teeth performed using a dental operating microscope at 8×-16× magnification.

SUMMARY:
The aim of this observational study is to compare the treatment durations of different stages of routine root canal therapy performed on maxillary molar teeth using direct vision, magnification loupes, and a dental operating microscope.

The primary question the study seeks to answer is whether there is a significant difference in the duration of endodontic procedures performed under different magnification techniques.

Patients indicated for root canal treatment in their maxillary first molar teeth will receive standard root canal therapy in accordance with routine clinical protocols. The duration of each procedural step will be recorded and subsequently compared among the three magnification methods.

DETAILED DESCRIPTION:
In this observational study, routine root canal treatment procedures will be performed in accordance with standard endodontic protocols on patients who applied to the Department of Endodontics, Faculty of Dentistry, Uşak University, and were indicated for root canal treatment on their maxillary first molar teeth.

1. The treatment procedures consist of seven main stages:
2. Preparation of the access cavity
3. Determination of the working length
4. Shaping of the root canals
5. Detection and shaping of the MB2 canal
6. Final irrigation and passive ultrasonic activation
7. Root canal filling

Application of the coronal restoration

All steps will be carried out according to standard clinical endodontic protocols under rubber dam isolation. The duration of each stage will be recorded individually.

Participants will be divided into three groups based on the magnification technique used during treatment:

Group 1: Treatments performed under direct vision

Group 2: Treatments performed using dental loupes

Group 3: Treatments performed using a dental operating microscope

All procedures in each group will follow the same standardized root canal treatment protocol, differing only in the magnification technique employed.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring root canal treatment of the maxillary first molar tooth

Exclusion Criteria:

* Previous root canal treatment on the maxillary first molar tooth
* Presence of fracture or crack in the maxillary first molar tooth
* Lack of indication for completing treatment in a single session
* Patient refusal to continue treatment during the procedure
* Indication for extraction due to complications during treatment
* Teeth indicated for fiber post restoration due to excessive material loss

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the Department of Endodontics, Faculty of Dentistry, Uşak University, who required root canal treatment of maxillary first molar teeth
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Duration of each procedural step in endodontic treatment | From the start of access cavity preparation to the completion of coronal restoration during a single treatment visit (approximately 35-120 minutes).
  The duration (in seconds) of each of seven key procedural stages performed during routine root canal treatment on maxillary first molar teeth:
  1. Access cavity preparation
  2. Working length determination
  3. Canal shaping
  4. MB2 canal detection and shaping
  5. Final irrigation and passive ultrasonic activation
  6. Root canal filling
  7. Coronal restoration
  Each stage was timed separately for three groups (direct vision, dental loupes, and dental operating microscope) to compare the effect of different magnification techniques on working efficiency.

SECONDARY OUTCOMES:
Presence of MB2 canal according to magnification technique | Baseline (at the time of canal orifice identification)
  The presence or absence of a second mesiobuccal (MB2) canal in maxillary first molar teeth will be recorded for each magnification group (direct vision, dental loupes, and dental operating microscope). The association between the magnification method and MB2 canal detection will be evaluated using the Chi-square test (Monte Carlo simulation).

CONTACTS AND LOCATIONS:
Overall Officials: Oğuz Tavşan, Assistant Professor, Principal Investigator — Uşak University Faculty of Dentistry, Department of Endodontics; Tuğçe N Çağlar, Research Assistant, Study Director — Uşak University Faculty of Dentistry, Department of Endodontics
Locations (1):
- Uşak University Faculty of Dentistry, Department of Endodontics, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data collected in this study will not be shared with other researchers. Data will be used only for academic purposes within the scope of the thesis and institutional ethics approval.

REFERENCES:
- [Background] Buhrley LJ, Barrows MJ, BeGole EA, Wenckus CS. Effect of magnification on locating the MB2 canal in maxillary molars. J Endod. 2002 Apr;28(4):324-7. doi: 10.1097/00004770-200204000-00016. PMID 12043874
- [Background] Malpas JS, Freeman JE. Blood and neoplastic diseases. Solid tumours in children. Br Med J. 1974 Dec 21;4(5946):710-3. doi: 10.1136/bmj.4.5946.710. No abstract available. PMID 4374292